CLINICAL TRIAL: NCT03830398
Title: Comparison of Paracetamol and Dexketoprofen Trometamol on Headache Treatment After Electroconvulsive Treatment
Brief Title: Comparison of Drugs on Headache Treatment After ECT Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Onur Koyuncu, Assoc.Prof.MD, Mustafa Kemal University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018/171
Record Dates: First submitted 2019-01-15; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Each drug for one week
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Paracetamol (Active Comparator): Parol group: intravenous infusion in 30 min Generic name: Parol Dosage form: intravenous Dosage: 1 gr Frequency: preop one dose only Duration: For one week
  Interventions: Drug: Paracetamol
- Deksketoprofen trometamol (Active Comparator): Sertofen group: intravenous infusion in 30 min Generic name: Sertofen Dosage form: intravenous Dosage: 50 mg Frequency: preop one dose only Duration: For one week
  Interventions: Drug: Deksketoprofen trometamol
- Placebo (Placebo Comparator): Placebo group: intravenous infusion in 30 min Generic name: Serum physiologic Dosage form: intravenous Dosage: 100 ml Frequency: preop one dose only Duration: For one week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol — The investigators apply paracetamol during a week in preoperative room 45 min before ECT
  Other Names: Parol
  Arms: Paracetamol
Drug: Deksketoprofen trometamol — The investigators apply paracetamol during a week in preoperative room 45 min before ECT
  Other Names: Sertofen
  Arms: Deksketoprofen trometamol
Drug: Placebo — The investigators apply placebo during a week in preoperative room 45 min before ECT
  Other Names: Serum Physiologic
  Arms: Placebo

SUMMARY:
Electroconvulsive treatment (ECT) is still actual for treatment of psychiatric symptoms. Headache is a very common symptom after this application. The investigators compare the effect of two different drugs for the treatment of headache after ECT.

DETAILED DESCRIPTION:
Electroconvulsive treatment (ECT) is used as an alternative application instead of drug therapy for psychiatric symptoms. ECT application is repeated 8-12 times according to the treatment of the patient. This treatment is done in 2 or 3 days intervals. The most adverse effects of ECT are headache, memory disorders, myalgia, nausea and vomiting, cardiovascular problems. The most common seen adverse effect is headache with approximately 60% incidence. The main drugs used for the treatment of headache related to ECT are NSAIs and paracetamol. The aim of the current study is to compare the effect of paracetamol and dexketoprofen trometamol on headache treatment after ECT.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were admitted for ECT and gave informed written consent were included in the study.

Exclusion Criteria:

* Exclusion criteria included patients who gave a history of allergy to acetaminophen, lacked capacity to give informed consent and developed complications such as delirium following ECT.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Headache (Visual Analogue Scale 0-10) | Postoperative 2. hour, 4. hour, 6. hour (up to six hours after intervention)
  Headache (VAS) change is being assessed in three different time frames after ECT

SECONDARY OUTCOMES:
Additive analgesic-antiemetic consumption | Postoperative 2. hour, 4. hour, 6. hour (up to six hours after intervention)
  If VAS ≥ 4, then diclofenac sodium im is given- If nausea-vomiting occurs, ondansetrone 4mg iv is given.The numbers of given drugs will be recorded in each interval.
Adverse effects (Nausea-Vomiting, bradycardia, hypotension) | Postoperative 2. hour, 4. hour, 6. hour (up to six hours after intervention)
  Number of adverse efffects will be recorded in each interval.

CONTACTS AND LOCATIONS:
Overall Officials: Onur Koyuncu, Asc.Prof, Principal Investigator — Mustafa Kemal Univ.; Sedat Hakimoglu, Asc.Prof, Study Chair — Mustafa Kemal Univ.; Senem Urfalı, Ast.Prof, Study Director — Mustafa Kemal Univ.; Sumeyra Yesil, Resident, Principal Investigator — Mustafa Kemal Univ.
Locations (1):
- Mustafa Kemal University Medicine Faculty Anesthesiology Department, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Isuru A, Rodrigo A, Wijesinghe C, Ediriweera D, Premadasa S, Wijesekara C, Kuruppuarachchi L. A randomized, double-blind, placebo-controlled trial on the role of preemptive analgesia with acetaminophen [paracetamol] in reducing headache following electroconvulsive therapy [ECT]. BMC Psychiatry. 2017 Jul 28;17(1):275. doi: 10.1186/s12888-017-1444-6. PMID 28754173